CLINICAL TRIAL: NCT04468685
Title: Efficacy of Intraperitoneal Ondansetron Administration on Pain Relief After Laparoscopic Cholecystectomy
Brief Title: Ondansetron Effect on Pain Relief After Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, Doaa abdelaziz, Lecturer of clinical pharmacy, National Hepatology & Tropical Medicine Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-2020
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis | interventions — Ondansetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ondansetron (Experimental): Ondansetron intraperitoneal in the gall bladder bed
  Interventions: Drug: Ondansetron
- Saline (Placebo Comparator): Normal saline intraperitoneal in the gall bladder bed
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ondansetron — Interperitoneal administration in the gall bladder bed
  Arms: Ondansetron
Drug: Normal saline — Interperitoneal administration in the gall bladder bed
  Arms: Saline

SUMMARY:
Laparoscopic cholecystectomy (LC) is an easy procedure characterized by its minimal invasiveness, less post-operative pain and early recovery when compared to the open conventional cholecystectomy. However, patients who have undergone LC still complain of postoperative pain. It has been reported that ondansetron produces numbness when injected under the skin and has local anesthetic effect that is 15 times more potent than lidocaine the most widely used local anesthetic and probably explains its antiemetic action. It possesses anti-inflammatory, anesthetic, and analgesic properties by its multifaceted actions as a 5-HT3 receptor antagonist, a Na channel blocker, and a mu-opioid agonist which may have a potential role in decreasing pain. The study aimed to demonstrate the effectiveness of IP administration of ondansetron on pain management post LC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo elective LC

Exclusion Criteria:

* Patients undergoing chronic pain treatment
* Previous allergic response to local anesthetics or 5-HT3 receptor antagonists
* Patients who received analgesics or sedatives 24 h before scheduled surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
change in postoperative pain between the two groups using visual analogue score (VAS) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The National Hepatology and Tropical Research medicine institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No